CLINICAL TRIAL: NCT01601678
Title: Endoscopic Versus Laparoscopic Myotomy for Treatment of Idiopathic Achalasia: A Randomized, Controlled Trial
Brief Title: Endoscopic Versus Laparoscopic Myotomy for Treatment of Idiopathic Achalasia
Acronym: POEMrct
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Karolinska University Hospital (Other); University Hospital Prague (IKEM), Prague, Czech Republic (Unknown); Universitaire Ziekenhuizen KU Leuven (Other); Istituto Clinico Humanitas (Other); Wuerzburg University Hospital (Other); University Hospital Augsburg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Rösch, Prof. Dr. Thomas Roesch, Universitätsklinikum Hamburg-Eppendorf, Endoscopy department, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POEM vs. LHM; PV 4133 (Registry Identifier: Hamburg Chamber of Physicians)
Record Dates: First submitted 2012-05-15; First posted 2012-05-18 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Achalasia
Keywords: Achalasia; Heller Myotomy; Dysphagia; Peroral Endoscopic Myotomy; LHM; POEM
MeSH Terms: conditions — Esophageal Achalasia; Deglutition Disorders | interventions — Heller Myotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peroral Endoscopic Myotomy POEM (Active Comparator): Patients with Achalasia, designated to receive a myotomy of the lower esophageal sphincter, who have been randomised into the POEM therapy group
  Interventions: Procedure: Peroral Endoscopic Myotomy (POEM)
- Laparoscopic Heller Myotomy LHM (Active Comparator): Patients with Achalasia, designated to receive a myotomy of the lower esophageal sphincter, who have been randomised into the LHM therapy group.
  Interventions: Procedure: Laparoscopic Heller Myotomy (LHM)

INTERVENTIONS:
Procedure: Peroral Endoscopic Myotomy (POEM) — After lavage, measure gastro-esophageal junction (GEJ) in cm from mouth piece. Determine entry point 12-14cm above GEJ at the lesser curvature site, inject 10ml coloured saline, create entry point. Advance endoscope into the submucosa, dissect the submucosal tunnel up to 2-3cm into the cardia. Dissect the submucosa close to the muscularis and check endoluminally for the direction of the lesser curvature, sufficient extension onto the cardia and mucosal integrity. After tunnel completion flush with gentamycin and saline. Start myotomy from proximally to distally starting 4-5cm below the mucosal entry site; the inner circular muscle layer should be fully dissected especially at the cardia for good symptomatic results. It is vital that the mucosa of the tubular esophagus remains intact. Extend myotomy at least 2cm onto the cardia. After completion check for mucosal integrity and opening of the distal esophageal sphincter. Close the entry point with clips from distal to proximal.
  Arms: Peroral Endoscopic Myotomy POEM
Procedure: Laparoscopic Heller Myotomy (LHM) — Use five trocar technique with patient in the French position as for laparoscopic anti-reflux procedures. Establish 12-15 mm Hg pneumoperitoneum. Use left paramedian trocar for camera, two lateral trocars for elevating liver and retraction of stomach and two trocars for dissection and suturing. Use of robotic surgery devices is allowed. Divide phrenoesophageal ligament starting on the right and mobilize distal esophagus on the lateral and anterior side. Identify and spare anterior vagal nerve. Perform myotomy by dividing both muscle-layers extending at least 6 cm above gastroesophageal junction and at least 2-3 cm inferiorly over stomach. Perform extent downwards after dividing epiphrenic fat pad overlying cardia. Measure myotomy length. Peroperative endoscopy check is advisable. Perform anterior fundoplication according to Dor. Only if necessary mobilize fundus of the stomach by dividing short gastric vessels. Suture fundus to both cut edges of myotomy, using non-resorbable material.
  Arms: Laparoscopic Heller Myotomy LHM

SUMMARY:
Achalasia is a rare neurodegenerative esophageal motility disorder characterized by incomplete lower esophageal sphincter (LES) relaxation, increased LES tone, and aperistalsis of the esophagus leading to dysphagia, regurgitation, and chest pain. therapies for achalasia consist of endoscopic balloon dilatation (EBD) and botulinum toxin injection (EBTI), or surgical Treatment via i Heller Myotomy; surgery is nowadays mostly performed via the laparoscopic approach. Surgical therapy demonstrated superior treatment efficacy compared to EBD and EBTI. Recently, an endoscopic means to perform myotomy via a submucosal tunnel has been developed, namely PerOral Endoscopic Myotomy (POEM). Uncontrolled studies have indicated a symptomatic success rate of >90% for POEM in short term follow-ups.The aim of this study is to compare short and long-term feasibility, safety and efficacy of endoscopic (POEM) with laparoscopic myotomy (Heller myotomy) in the treatment of achalasia.

DETAILED DESCRIPTION:
Achalasia is considered a primary esophageal motility disorder which is defined as an insufficient relaxation of the lower esophageal sphincter. Incomplete lower esophageal sphincter (LES) relaxation, increased LES tone, and aperistalsis of the esophagus are characteristics of achalasia. Incidence peaks between ages 20 to 40. The most commonly reported symptoms are dysphagia (both for solids and liquids), regurgitation, and chest pain. The diagnosis is established with esophageal manometry and barium swallow radiographic studies and also with endoscopy being performed to exclude neoplastic or inflammatory diseases. Endoscopic therapies consist of either balloon dilatation (EBD) or Botulinum toxin injection (EBTI). The surgical treatment for achalasia is Heller Myotomy, nowadays almost exclusively performed laparoscopically.Superior to EBD and EBTI, surgical myotomy has shown sustained therapeutic efficacy in approximately 90% of patients which may be especially relevant for young patients with achalasia.

Recently an endoscopic technique to create myotomy via a submucosal tunnel has been developed, named PerOral Endoscopic Myotomy (POEM). The technique was first reported by Pasricha et al. in a porcine study, and Inoue et al. later reported the first clinical results in achalasia patients which showed significantly reduced dysphagia symptom scores and decreased resting lower esophageal sphincter (LES) pressures in 17 patients with a mean follow-up of 5 months . No serious complications related to POEM were encountered in this initial single-center trial. Several smaller pilot studies from Asia, Europe and USA have replicated the promising results regarding feasibility, safety and short-term efficacy,leading us to hope for a similar success rate along with reduced patient discomfort At present, POEM has the potential to be the first scarless flexible endosurgical intervention to become an established clinical treatment.The technique uses a submucosal esophageal tunnel through which a distal esophageal myotomy down to the proximal stomach is performed. For POEM to be integrated into clinical routine, comparative data regarding safety and efficacy are necessary.Our study group intends to compare safety and long-term efficacy of POEM to laparoscopic Heller myotomy, the current gold-Standard, in a non-inferiority design.

Patients with symptomatic achalasia and medical indication for interventional therapy will be randomized to either POEM therapy or standard laparoscopic Heller myotomy (with anti-reflux procedure)(LHM). They will be followed up closely in a defined time pattern evolving individual life quality and achalasia scores as well as clinical scores and diagnostics over a period of 5 years.

Due to considerations concerning the comparability to other achalsia Trials (Boeckxstaens,NEJM 2011), in November 2012 primary outcome has been changed to Eckardt Score instead of lower sphicter pressure. Amendment was done before patient inclusion started. Sample size was not affected by amendment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic achalasia with an Eckardt score of > 3 and pre-op barium swallow, manometry and esophagogastroduodenoscopy consistent with the diagnosis
* Persons of age > 18 years with medical indication for surgical myotomy or EBD
* Signed written Informed Consent

Exclusion Criteria:

* Patients with previous surgery of the stomach or esophagus
* Patients with known coagulopathy
* Previous surgical achalasia treatment
* Patients with liver cirrhosis and/or esophageal varices
* Active esophagitis
* Eosinophilic esophagitis
* Barrett's esophagus
* Pregnancy
* Stricture of the esophagus
* Malignant or premalignant esophageal lesion
* Severe Candida esophagitis
* Hiatal hernia > 1cm
* Extensive tortuous dilatation (>7cm luminal diameter, S shape) of the esophagus
* Advanced malignant tumor with prognosis < 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Eckhard symptom scores | 2 years after treatment
  Achalasia symptom questionnaire to evaluate individual therapy success, range from 0 (no Achalasia symptoms) to 12 (full symptom range), treatment success is defined as an Eckardt Score ≤ 3

SECONDARY OUTCOMES:
Eckhard symptom scores | before,and 3 and 6 months, 1,3 and 5 years past procedure
  Achalasia symptom questionnaire to evaluate individual therapy success, range from 0 (no Achalasia symptoms) to 12 (full symptom range)
Treatment success rates | 3 and 6 months, and 1, 3, and 5 years post procedure
  success rates result from Eckardt Scores
Manometry data | before, and 3 months, and 2 and 5 years post procedure
  Achalasia subtypes (before treatment) and assessment of lower esophagus sphincter function
Reflux score (clinical DeMeester score) | before, and 3 and 6 months, and 1, 2, 3, and 5 years post procedure
  clinical DeMeester Reflux questionnaire to evaluate therapeutic side effects, range from 0 (no Reflux symptoms) to 6 (full symptom range).
Reflux symptoms | before, and 3 and 6 months, and 1, 2, 3, and 5 years post procedure
  List of side effects due to reflux past POEM as short term and long term outcomes
pH metry | 3 months and 2 and 5 years after therapy
  pH metry data after therapy
Adverse Events | Baseline to five years past procedure
  complication rate (Adverse Events (AE) and Serious Adverse Events (SAE))
Quality of Life index | before, and 3 months, and 2 and 5 years post procedure
  Life quality assessment (gastrointestinal LQ index by Eypasch, Wood-Dauphinee and Troidl) for individual success Evaluation (GIQLI), Best outcome score is 144.
EGD findings | 3 months and (optional) 2 and 5 years after therapy
  EGD findings to evaluate reflux effects after therapy
CRP lab values | day before procedure to day after procedure
  CRP values measured in mg/l (milligrams per litre) pre and post procedure
Hb lab values | day before procedure to day after procedure
  Hemoglobin values measured in g/dl (grams per decilitre) pre and post procedure
Leucocyte lab values | day before procedure to day after procedure
  Leucocyte values measured in billions per litre pre and post procedure, number of days of hospitalisation, myotomy length, duration of procedure
number of days of hospitalisation | through inhouse stay after procedure, an average of 2-7 days
  inhouse stay after procedure
myotomy length | day of procedure
  myotomy length in cm
duration of procedure | day of procedure
  duration of procedure in minutes
Therapy failures | from procedure to 5 years after procedure
  number of therapy failures
Retreatments | from procedure to 5 years after procedure
  number and kinds of retreatments

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Roesch, Prof., Study Director — Interdisciplinary Endoscopy Department and Clinic, University Hospital Hamburg-Eppendorf, Germany; Paul Fockens, Prof., Principal Investigator — Department of Gastroenterology and Hepatology, Academic Medical Center, Amsterdam; Netherlands; Bengt Håkanson, Prof., Principal Investigator — Department of Surgery, Karolinska University Hospital, Stockholm, Sweden; Guy Boeckxstaens, Prof., Principal Investigator — Universitaire Ziekenhuizen KU Leuven; C.T. Germer, Prof., Principal Investigator — Wuerzburg University Hospital; Riccardo Repici, Prof., Principal Investigator — Istituto Clinico Humanitas, Rozzano, Italy; Uberto Fumagalli, Prof., Principal Investigator — Istituto Clinico Humanitas, Rozzano, Italy; Julius Spicak, Prof., Principal Investigator — University Hospital Prague, Prague, Czech Republic; Helmut Messmann, Prof., Principal Investigator — Department for Internal Medicine III, Klinikum Augsburg, Germany
Locations (8):
- University Hospital Leuven, Leuven, Belgium
- University Hospital Prague (IKEM), Prague, Czechia
- Germany (3):
  - Klinikum Augsburg,Klinik für Innere Medizin III, Augsburg
  - Universitätsklinikum Eppendorf, Hamburg
  - University Hospital Würzburg, Würzburg
- Istituto Clinico Humanitas, Rozzano, Italy
- Academic Medical Center, Amsterdam, Netherlands
- Ersta Hospital and Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campos GM, Vittinghoff E, Rabl C, Takata M, Gadenstatter M, Lin F, Ciovica R. Endoscopic and surgical treatments for achalasia: a systematic review and meta-analysis. Ann Surg. 2009 Jan;249(1):45-57. doi: 10.1097/SLA.0b013e31818e43ab. PMID 19106675
- [Background] von Rahden BH, Germer CT. [Laparoscopic myotomy for achalasia is clearly superior to the endoscopic treatment]. Chirurg. 2010 Jan;81(1):69-70. doi: 10.1007/s00104-009-1840-7. No abstract available. German. PMID 19940967
- [Background] Rebecchi F, Giaccone C, Farinella E, Campaci R, Morino M. Randomized controlled trial of laparoscopic Heller myotomy plus Dor fundoplication versus Nissen fundoplication for achalasia: long-term results. Ann Surg. 2008 Dec;248(6):1023-30. doi: 10.1097/SLA.0b013e318190a776. PMID 19092347
- [Background] Ortiz A, de Haro LF, Parrilla P, Lage A, Perez D, Munitiz V, Ruiz D, Molina J. Very long-term objective evaluation of heller myotomy plus posterior partial fundoplication in patients with achalasia of the cardia. Ann Surg. 2008 Feb;247(2):258-64. doi: 10.1097/SLA.0b013e318159d7dd. PMID 18216530
- [Background] Perretta S, Dallemagne B, Allemann P, Marescaux J. Multimedia manuscript. Heller myotomy and intraluminal fundoplication: a NOTES technique. Surg Endosc. 2010 Nov;24(11):2903. doi: 10.1007/s00464-010-1073-3. Epub 2010 Apr 29. PMID 20428893
- [Background] Pasricha PJ, Hawari R, Ahmed I, Chen J, Cotton PB, Hawes RH, Kalloo AN, Kantsevoy SV, Gostout CJ. Submucosal endoscopic esophageal myotomy: a novel experimental approach for the treatment of achalasia. Endoscopy. 2007 Sep;39(9):761-4. doi: 10.1055/s-2007-966764. PMID 17703382
- [Background] Inoue H, Minami H, Kobayashi Y, Sato Y, Kaga M, Suzuki M, Satodate H, Odaka N, Itoh H, Kudo S. Peroral endoscopic myotomy (POEM) for esophageal achalasia. Endoscopy. 2010 Apr;42(4):265-71. doi: 10.1055/s-0029-1244080. Epub 2010 Mar 30. PMID 20354937
- [Background] von Renteln D, Inoue H, Minami H, Werner YB, Pace A, Kersten JF, Much CC, Schachschal G, Mann O, Keller J, Fuchs KH, Rosch T. Peroral endoscopic myotomy for the treatment of achalasia: a prospective single center study. Am J Gastroenterol. 2012 Mar;107(3):411-7. doi: 10.1038/ajg.2011.388. Epub 2011 Nov 8. PMID 22068665
- [Background] Swanstrom LL, Rieder E, Dunst CM. A stepwise approach and early clinical experience in peroral endoscopic myotomy for the treatment of achalasia and esophageal motility disorders. J Am Coll Surg. 2011 Dec;213(6):751-6. doi: 10.1016/j.jamcollsurg.2011.09.001. Epub 2011 Oct 13. PMID 21996484
- [Background] Boeckxstaens GE, Annese V, des Varannes SB, Chaussade S, Costantini M, Cuttitta A, Elizalde JI, Fumagalli U, Gaudric M, Rohof WO, Smout AJ, Tack J, Zwinderman AH, Zaninotto G, Busch OR; European Achalasia Trial Investigators. Pneumatic dilation versus laparoscopic Heller's myotomy for idiopathic achalasia. N Engl J Med. 2011 May 12;364(19):1807-16. doi: 10.1056/NEJMoa1010502. PMID 21561346
- [Background] ZHOU PH, CAI MY, YAO LQ, ZHONG YS, REN Z, XU MD, CHEN WF, QIN XY. [Peroral endoscopic myotomy for esophageal achalasia: report of 42 cases]. Zhonghua Wei Chang Wai Ke Za Zhi. 2011 Sep;14(9):705-8. Chinese. PMID 21948538
- [Background] Smith CD, Stival A, Howell DL, Swafford V. Endoscopic therapy for achalasia before Heller myotomy results in worse outcomes than heller myotomy alone. Ann Surg. 2006 May;243(5):579-84; discussion 584-6. doi: 10.1097/01.sla.0000217524.75529.2d. PMID 16632991
- [Derived] Hugova K, Mares J, Hakanson B, Repici A, von Rahden BHA, Bredenoord AJ, Bisschops R, Messmann H, Ruppenthal T, Mann O, Izbicki J, Harustiak T, Fumagalli Romario U, Rosati R, Germer CT, Schijven M, Emmermann A, von Renteln D, Dautel S, Fockens P, Boeckxstaens G, Rosch T, Martinek J, Werner YB. Per-oral endoscopic myotomy versus laparoscopic Heller's myotomy plus Dor fundoplication in patients with idiopathic achalasia: 5-year follow-up of a multicentre, randomised, open-label, non-inferiority trial. Lancet Gastroenterol Hepatol. 2025 May;10(5):431-441. doi: 10.1016/S2468-1253(25)00012-3. Epub 2025 Mar 17. PMID 40112837
- [Derived] Werner YB, Hakanson B, Martinek J, Repici A, von Rahden BHA, Bredenoord AJ, Bisschops R, Messmann H, Vollberg MC, Noder T, Kersten JF, Mann O, Izbicki J, Pazdro A, Fumagalli U, Rosati R, Germer CT, Schijven MP, Emmermann A, von Renteln D, Fockens P, Boeckxstaens G, Rosch T. Endoscopic or Surgical Myotomy in Patients with Idiopathic Achalasia. N Engl J Med. 2019 Dec 5;381(23):2219-2229. doi: 10.1056/NEJMoa1905380. PMID 31800987